CLINICAL TRIAL: NCT03786770
Title: A Phase 2a, Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Efficacy and Safety of DaxibotulinumtoxinA (DAXI) for Injection for the Treatment of Dynamic Forehead Lines (Frontalis) Following Glabellar Line Injections
Brief Title: Efficacy and Safety of DaxibotulinumtoxinA (DAXI) for Injection for Treatment of Forehead Lines (Frontalis)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1820202
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Frown Lines
Keywords: Forehead Lines; Glabellar Lines; Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Dose A (Experimental): DAXI for injection for the treatment of Forehead Lines (FHL) and Glabellar Lines (GL)
  Interventions: Biological: DaxibotulinumtoxinA for injection
- Cohort 2: Dose B (Experimental): DAXI for injection for the treatment of Forehead Lines (FHL) and Glabellar Lines (GL)
  Interventions: Biological: DaxibotulinumtoxinA for injection
- Cohort 3: Dose C (Experimental): DAXI for injection for the treatment of Forehead Lines (FHL) and Glabellar Lines (GL)
  Interventions: Biological: DaxibotulinumtoxinA for injection
- Cohort 4: Dose D (Experimental): DAXI for injection for the treatment of Forehead Lines (FHL) and Glabellar Lines (GL)
  Interventions: Biological: DaxibotulinumtoxinA for injection

INTERVENTIONS:
Biological: DaxibotulinumtoxinA for injection — Intramuscular injection

SUMMARY:
This is a phase 2a, multicenter, open-label, dose-escalation study to evaluate treatment of moderate or severe dynamic forehead lines (FHL) (frontalis) in conjunction with treatment of the glabellar complex.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent consistent with International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines and local laws, including authorization to release health information, signed prior to any study procedures being performed
* Be outpatient, male or female subjects, in good general health, 18-65 years of age
* Have a score of moderate (2) or severe (3) FHL during maximum contraction (eyebrow elevation) as assessed by the Investigator Global Assessment Forehead Wrinkle Severity (IGA-FHWS)
* Have a score of moderate (2) or severe (3) FHL during maximum contraction (eyebrow elevation) as assessed by the Patient Forehead Wrinkle Severity (PFHWS)
* Have a score of moderate (2) or severe (3) GL during maximum frown based on the Investigator Global Assessment Frown Wrinkle Severity (IGA-FWS) scale
* Have a score of moderate (2) or severe (3) on GL during maximum frown as assessed by the Patient Frown Wrinkle Severity (PFWS)
* Be willing to refrain from receiving facial fillers, laser treatments, use of any product that affects skin remodeling, or a product that may cause an active dermal response in the treatment areas (e.g., above the inferior orbital rim) from screening through the end of the study
* Able to understand the requirements of the study and be willing and able to follow all study procedures, attend all scheduled visits, and successfully complete the study.

Exclusion Criteria:

* Active skin disease, infections, or inflammation at the injection sites
* Plans to receive botulinum toxin type A anywhere in the face (other than study treatment) from screening through the end of the study
* History of clinically significant bleeding disorders
* Non-ablative laser or light treatments, microdermabrasion, or chemical peels (medium depth or deeper, for example trichloroacetic acid (TCA) or phenol) in the treatment areas within 3 months before enrollment through the end of the study
* Clinically significant laboratory values at screening that may interfere with a subject's ability to complete the study as determined by the investigator
* History of upper or lower lid blepharoplasty or brow lift
* Prior periorbital or forehead surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Boca Raton site, Boca Raton, Florida
  - Coral Gables site, Coral Gables, Florida
- Canada (2):
  - Toronto, Ontario site, Toronto, Ontario
  - Woodbridge, Ontario site, Woodbridge, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: DAXI 40 U GL / 12 U FHL: DAXI for injection for the treatment of Forehead Lines (FHL) with 12 U and Glabellar Lines (GL) with 40 U
- Cohort 2: DAXI 40 U GL / 18 U FHL: DAXI for injection for the treatment of Forehead Lines (FHL) with 18 U and Glabellar Lines (GL) with 40 U
- Cohort 3: DAXI 40 U GL / 24 U FHL: DAXI for injection for the treatment of Forehead Lines (FHL) with 24 U and Glabellar Lines (GL) with 40 U
- Cohort 4: DAXI 40 U GL / 30 U FHL: DAXI for injection for the treatment of Forehead Lines (FHL) with 30 U and Glabellar Lines (GL) with 40 U
Period: Overall Study
Arm/Group | Cohort 1: DAXI 40 U GL / 12 U FHL | Cohort 2: DAXI 40 U GL / 18 U FHL | Cohort 3: DAXI 40 U GL / 24 U FHL | Cohort 4: DAXI 40 U GL / 30 U FHL
Started | 14 | 15 | 16 | 16
Completed | 13 | 15 | 16 | 16
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: DAXI 40 U GL / 12 U FHL | Cohort 2: DAXI 40 U GL / 18 U FHL | Cohort 3: DAXI 40 U GL / 24 U FHL | Cohort 4: DAXI 40 U GL / 30 U FHL | Total
Number analyzed (Participants) | 14 | 15 | 16 | 16 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 16 | 15 | 60
  >=65 years | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 49 [37 to 62] | 48.1 [34 to 60] | 47.8 [26 to 62] | 45.6 [28 to 65] | 47.6 [26 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 15 | 15 | 54
  Male | 4 | 1 | 1 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 14 | 15 | 15 | 15 | 59
  Race: Black/African American | 0 | 0 | 1 | 0 | 1
  Race: Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With None or Mild in FHL Severity at Maximum Eyebrow Elevation
Description: Percentage of subjects achieving a score of 0 or 1 (none or mild) in FHL severity at maximum eyebrow elevation at 4 weeks after FHL treatment (Week 6) on the 4-point Investigator Global Assessment Forehead Wrinkle Severity (IGA-FHWS) scale where 0 indicates the lowest severity and 3 indicates the highest severity.
Time Frame: Week 4 After FHL Treatment
Population: The FHL-evaluable population
Measure: Number; unit: percentage of subjects
Arm/Group | Cohort 1: DAXI 40 U GL / 12 U FHL | Cohort 2: DAXI 40 U GL / 18 U FHL | Cohort 3: DAXI 40 U GL / 24 U FHL | Cohort 4: DAXI 40 U GL / 30 U FHL
Number analyzed (Participants) | 14 | 15 | 16 | 15
percentage of subjects | 85.7 | 86.7 | 93.8 | 100

ADVERSE EVENTS:
Time Frame: The adverse events were collected throughout the entire study, up to 36 weeks after FHL treatment (total of 38 weeks).
Description: The Safety Population includes all subjects who received at least 1 study treatment injection and was used to assess AEs and SAEs
Arm/Group | Cohort 1: DAXI 40 U GL / 12 U FHL | Cohort 2: DAXI 40 U GL / 18 U FHL | Cohort 3: DAXI 40 U GL / 24 U FHL | Cohort 4: DAXI 40 U GL / 30 U FHL
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 5/14 | 5/15 | 5/16 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: DAXI 40 U GL / 12 U FHL (N=14) | Cohort 2: DAXI 40 U GL / 18 U FHL (N=15) | Cohort 3: DAXI 40 U GL / 24 U FHL (N=16) | Cohort 4: DAXI 40 U GL / 30 U FHL (N=16)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 4 (6) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 1 (1) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Center and/or Investigator shall submit to Revance a copy of the proposed publication at least sixty (60) days prior to the submission thereof for publication or disclosure to a third party: (i)to provide Revance with the opportunity to review and comment on the contents thereof, (ii)to identify any Confidential Information to be deleted from the proposed publication or disclosure, and (iii)or delay the publication or disclosure 90 days to allow Revance to pursue patent protections.

DOCUMENTS (2):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT03786770/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03786770/SAP_001.pdf